CLINICAL TRIAL: NCT04119843
Title: A Multicenter, Open-label Study to Evaluate the Safety and Diagnostic Efficacy of Mangoral in Patients With Known or Suspected Focal Liver Lesions and Severe Renal Impairment
Brief Title: Safety and Diagnostic Efficacy of Mangoral in Participants With Focal Liver Lesions and Reduced Kidney Function
Acronym: SPARKLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascelia Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ASC-Man-P016; 11-3429 (Other: FDA Orphan Designation Request)
Record Dates: First submitted 2019-09-29; First posted 2019-10-08 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Known or Suspected Focal Liver Lesions; Severe Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — CMC-001

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, pivotal phase III study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mangoral (Experimental): All participants will receive a single dose of Mangoral (800 mg Manganese (II) chloride tetrahydrate [MnCl2 4H2O]).
  Interventions: Drug: Mangoral

INTERVENTIONS:
Drug: Mangoral — 800 mg manganese chloride [II] tetrahydrate, 500 mg L-alanine, and 800 IU vitamin D3
  Other Names: Orviglance; CMC-001; ACE-MBCA

SUMMARY:
The overall objective of this study is to evaluate the safety and diagnostic efficacy of Mangoral in liver MRI in participants with known or suspected focal liver lesions and severe renal impairment. The diagnostic efficacy of Mangoral will be assessed in terms of visualization of detected focal liver lesions in combined MRI (CMRI: combined Mangoral-enhanced and unenhanced MRI) compared to unenhanced MRI.

DETAILED DESCRIPTION:
The overall objective of this multicenter, open-label, study is to evaluate the safety and diagnostic efficacy of Mangoral in participants with known or suspected focal liver lesions and severe renal impairment. Study treatment is a single oral dose of Mangoral (800 mg manganese chloride [II] tetrahydrate, 500 mg L-alanine, and 800 IU vitamin D3). Adult male and female participants with severe renal impairment or acute kidney injury and who are being evaluated for known or suspected focal liver lesions will be included. Primary diagnostic efficacy in terms of visualization of detected lesions will be evaluated centrally by 3 independent readers. Study MRIs will also be evaluated by the on-site radiologists for the assessment of secondary objectives and for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 years and older.
* Known or suspected focal liver lesions based on medical history and previous laboratory and/or imaging examinations.
* Severe renal impairment (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m^2) based on medical history and previous laboratory examinations, at least once, within the last 3 months prior to the Baseline Visit, or participants with an increase in serum creatinine ≥ 0.3 mg/dL within 48 hours or ≥ 50% within 7 days prior to the Baseline Visit.

Exclusion Criteria:

* Participants with simple liver cysts only.
* Any investigational drug or device within 6 weeks prior to the Baseline Visit.
* Any magnetic resonance imaging (MRI) contrast media within 6 weeks prior to Baseline Visit or scheduled to receive any contrast medium before the last study visit.
* Participants with severe hepatic impairment (according to Child-Pugh score C).
* Participants scheduled for surgery before last study visit.
* Participants with encephalopathy / neurodegenerative or acute neurological disorders.
* Participants with hemochromatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hamm, MD, Principal Investigator — Charite Berlin, Dept. of Radiology
Locations (60):
- United States (14):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - University of California at Los Angeles Ronald Reagan Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Schiff Center for Liver Diseases, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - PanAmerican Clinical Research LLC, Brownsville, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Argentina (3):
  - Fundación Intecnus, Bariloche, Río Negro Province
  - Centro Rossi Body Imaging, Buenos Aires
  - Sanatorio Allende Nueva Córdoba, Córdoba
- Colombia (3):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Clínica Universitaria Colombia, Bogotá, Cundinamarca
  - Sociedad de Cirugía de Bogotá - Hospital de San José, Bogotá, Cundinamarca
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt Institut für Diagnostische und Interventionelle Radiologie, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Städtisches Klinikum KarlsruheDiagnostische und interventionelle Radiologie, Karlsruhe
  - Universitättsklinikum Schleswig-Holstein/Campus KielKlinik für Radiologie und Neuroradiologie, Kiel
  - Klinik und Poliklinik für Radiologie Klinikum der Universität München LMU Campus, Munich
  - Institut für Röntgendiagnostik, Regensburg
- Italy (8):
  - Azienda Socio Sanitaria Territoriale (ASST), Milan, Lombardy
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale del Mare, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Rome
  - Ospedale di Belcolle, Viterbo
- Mexico (3):
  - Panamerican Clinical Research - Cuernavaca Rio Mayo, Cuernavaca
  - Panamerican Clinical Research Mexico, Guadalajara
  - Panamerican Clinical Research - Querétaro Avenida Paseo de la República, Querétaro
- Poland (3):
  - Szpital Uniwersytecki nr 1 im. Dr A. Jurasza, Wydział Katedra i Zakład Radiologii i Diagnostyki Obrazowej, Bydgoszcz
  - Szpital Uniwersytecki w Krakowie Zakład Diagnostyki Obrazowej CUMRiK Ul, Krakow
  - EuroMedis Sp. z o.o., Szczecin
- Russia (13):
  - Altay Regional Oncology Dispencery, Barnaul
  - State Institution of Healthcare "Regional Oncology Dispensary", Irkutsk
  - Scientific and Research Institute of Oncology named after N.N. Blokhin, Moscow
  - A.V. Vishnevsky Institute of Surgery, Moscow
  - National Medical Research Radiology Center Named After Herzen, Moscow
  - JSC "Avicenna", Novosibirsk
  - State Institution of Healthcare of Omsk region, Omsk
  - SBIH of Pskov Regional Clinical Oncologic Dispensary, Pskov
  - LLC "Clinica YZI 4D", Pyatigorsk
  - N.N. Petrov Research Institute of Oncology, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution, Saint Petersburg
  - Smolensk Clinical Hospital, Smolensk
  - State Autonomous Healthcare Institution of the Tyumen Region, Tyumen
- Karolinska University Hospital Huddinge, Stockholm, Sweden
- Turkey (Türkiye) (5):
  - Ege University Medical Faculty Hospital, Bornova, İzmir
  - Erciyes University Medical Faculty Hospital, Melikgazi, Kayseri
  - Kocaeli University, İzmit, Kocaeli
  - Hacettepe University Medical Faculty Hospital, Ankara
  - İstanbul Üniversitesi - Istanbul Tıp Fakültesi, Istanbul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 87 participants were enrolled in 32 study sites in Europe, Asia, North America, and South America between February 2020 and February 2023.
Pre-assignment Details: The study consisted of:
  * Screening Period (Day -28 to Day -1)
  * Baseline Period (Day -1 to Day 0, i.e., within 24 hours of mangoral administration) providing a Baseline magnetic resonance imaging (MRI) using an unenhanced MRI examination of the liver
  * Day of MRI (Day 0) included intake of mangoral after a fast of at least 4 hours and a mangoral-enhanced liver MRI 4 [±1] hours after mangoral administration
  * Follow-up visits following contrast administration (up to Day 7).
Groups:
- Mangoral: All participants received a single oral dose of mangoral (800 mg manganese [II] chloride tetrahydrate [MnCl2 4H2O]). Mangoral is a novel manganese-based contrast agent for liver MRI.
  Unenhanced MRI of the liver was performed during the Baseline Period, i.e., either on the day prior to the mangoral-enhanced MRI or predose on the same day as the mangoral-enhanced MRI. Mangoral-enhanced MRI of the liver was performed 4 (±1) hours after investigational medicinal product (IMP) administration. Each unenhanced and each mangoral-enhanced liver MRI examination will consist of axial T1- and T2-weighted image sequences and a diffusion-weighted imaging (DWI) sequence.
Period: Overall Study
Arm/Group | Mangoral
Started | 87
Underwent Unenhanced MRI | 85
Underwent Mangoral-enhanced MRI | 85
Completed | 83
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants enrolled in the study (fulfil all inclusion criteria, but none of the exclusion criteria and have been included in the clinical study at Visit 2).
Groups:
- Mangoral: All participants received a single oral dose of mangoral (800 mg). Mangoral is a novel manganese-based contrast agent for liver MRI.
  Unenhanced MRI of the liver was performed during the Baseline Period, i.e., either on the day prior to the mangoral-enhanced MRI or predose on the same day as the mangoral-enhanced MRI. Mangoral-enhanced MRI of the liver was performed 4 (±1) hours after IMP administration. Each unenhanced and each mangoral-enhanced liver MRI examination will consist of axial T1- and T2-weighted image sequences and a DWI sequence.
Arm/Group | Mangoral
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28
  Black or African American | 5
  American Indian or Alaska Native | 1
  Other | 6
  Unknown or Not Reported | 47

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Endpoint: Lesion Border Delineation in Combined MRI Compared to Unenhanced MRI
Description: Visualization of focal liver lesions was measured by 2 co-primary variables: 'lesion border delineation' and 'lesion contrast' compared to liver background. Qualitative assessment determined on the 4-point scales for up to 15 lesions per participant. Each lesion was assessed for lesion border delineation from 1 (poor: lesion border is poorly distinct) to 4 (excellent: lesion border is sharply and clearly distinct). Central reading sessions were undertaken by 3 independent, blinded readers.
  The scores were calculated for each participant by summing the individual lesion scores and calculating the mean. The total score could range from 1 to 4 for each participant with higher scores representing a better outcome.
Time Frame: Unenhanced MRI: Baseline Period (Day -1 to Day 0); combined MRI: Baseline Period (Day -1 to Day 0) and 4 hours after mangoral administration on Day 0
Population: Full Analysis Set (FAS): All participants of the Safety Population who received the IMP and for whom the primary efficacy variable was assessable, i.e. all unenhanced / enhanced liver MRI images are assessable. The overall number of participants analyzed includes all participants that contributed data for the outcome measure. The number of participants analyzed per row includes only participants with matched lesions (detected and scored on both unenhanced MRI and combined MRI) by each reader.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unenhanced MRI: All participants undertook an unenhanced MRI examination of the liver during the Baseline Period (Day -1 to Day 0, i.e., within 24 hours of mangoral administration).
  Unenhanced MRI was defined as the reading of the pre-mangoral, unenhanced MRI only.
- Combined MRI: All participants undertook an unenhanced MRI examination of the liver during the Baseline Period (Day -1 to Day 0, i.e., within 24 hours of mangoral administration).
  On the day of MRI (Day 0), all participants received a single oral dose of mangoral (800 mg) after a fast of at least 4 hours and undertook a mangoral-enhanced MRI examination of the liver 4 [±1] hours after mangoral administration.
  Combined MRI was defined as the paired, simultaneous reading of both unenhanced and mangoral-enhanced MRIs.
Arm/Group | Unenhanced MRI | Combined MRI
Number analyzed (Participants) | 85 | 85
score on a scale
  Reader 1: number analyzed (Participants) | 61 | 61
  Reader 1 | 2.51 (0.815) | 3.46 (0.861)
  Reader 2: number analyzed (Participants) | 53 | 53
  Reader 2 | 3.00 (0.952) | 3.80 (0.607)
  Reader 3: number analyzed (Participants) | 61 | 61
  Reader 3 | 2.31 (0.847) | 2.97 (0.782)
Statistical Analysis 1: Comparison: Unenhanced MRI vs Combined MRI; Paired difference of combined MRI versus unenhanced MRI: Reader 1; Test type: Superiority — Reader success for the primary analysis was achieved if the reading results demonstrated superiority of combined MRI versus unenhanced MRI for both lesion border delineation and lesion contrast. The acceptance by two out of three readers was considered to be a successful demonstration of efficacy in the study; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [0.743 to 1.165], Standard Deviation 0.824 — Positive changes in lesion border delineation mean difference (combined MRI compared to unenhanced MRI) represents a better outcome
Statistical Analysis 2: Comparison: Unenhanced MRI vs Combined MRI; Paired difference of combined MRI versus unenhanced MRI: Reader 2; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [0.552 to 1.043], Standard Deviation 0.892 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Unenhanced MRI vs Combined MRI; Paired difference of combined MRI versus unenhanced MRI: Reader 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [0.494 to 0.813], Standard Deviation 0.622 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Co-primary Endpoint: Lesion Contrast in Combined MRI Compared to Unenhanced MRI
Description: Visualization of focal liver lesions was measured by 2 co-primary variables: 'lesion border delineation' and 'lesion contrast' compared to liver background. Qualitative assessment determined on the 4-point scales for up to 15 lesions per participant. Each lesion was assessed for lesion contrast from 1 (poor: difference in signal intensity between the lesion and the surrounding normal liver tissue is poor) to 4 (excellent: difference in signal intensity between the lesion and the surrounding liver is marked). Central reading sessions were undertaken by 3 independent, blinded readers.
  The scores were calculated for each participant by summing the individual lesion scores and calculating the mean. The total score could range from 1 to 4 for each participant with higher scores representing a better outcome.
Time Frame: as for outcome 1
Population: FAS: All participants of the Safety Population who received the IMP and for whom the primary efficacy variable was assessable, i.e. all unenhanced / enhanced liver MRI images are assessable. The overall number of participants analyzed includes all participants that contributed data for the outcome measure. The number of participants analyzed per row includes only participants with matched lesions (detected and scored on both unenhanced MRI and combined MRI) by each reader.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Combined MRI: All participants undertook an unenhanced MRI examination of the liver during the Baseline Period (Day -1 to Day 0, i.e., within 24 hours of mangoral administration).
  On the day of MRI (Day 0), all participants received a single oral dose of mangoral (800 mg) after a fast of at least 4 hours and undertook a mangoral-enhanced MRI examination of the liver (paired with unenhanced MRI; combined MRI) 4 [±1] hours after mangoral administration.
  Combined MRI was defined as the paired, simultaneous reading of both unenhanced and mangoral-enhanced MRIs.
Arm/Group | Unenhanced MRI | Combined MRI
Number analyzed (Participants) | 85 | 85
score on a scale
  Reader 1: number analyzed (Participants) | 61 | 61
  Reader 1 | 2.49 (0.813) | 3.47 (0.844)
  Reader 2: number analyzed (Participants) | 53 | 53
  Reader 2 | 2.84 (0.926) | 3.86 (0.417)
  Reader 3: number analyzed (Participants) | 61 | 61
  Reader 3 | 2.51 (0.919) | 3.33 (0.684)
Statistical Analysis 1: Comparison: Unenhanced MRI vs Combined MRI; Paired difference of combined MRI versus unenhanced MRI: Reader 1; Test type: Superiority — Reader success of the primary analysis was achieved if the reading results demonstrated superiority of combined MRI versus unenhanced MRI for both lesion border delineation and lesion contrast. The acceptance by two out of three readers was considered to be a successful demonstration of efficacy in the study; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [0.759 to 1.196], Standard Deviation 0.853 — Positive changes in lesion contrast mean difference (combined MRI compared to unenhanced MRI) represents a better outcome
Statistical Analysis 2: Comparison: Unenhanced MRI vs Combined MRI; Paired difference of combined MRI versus unenhanced MRI: Reader 2; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [0.766 to 1.267], Standard Deviation 0.909 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Unenhanced MRI vs Combined MRI; Paired difference of combined MRI versus unenhanced MRI: Reader 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [0.638 to 0.985], Standard Deviation 0.678 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Lesions Detected by Each MRI Method
Description: Assessments of unenhanced MRI, mangoral-enhanced MRI, and combined MRI for detection of lesions were undertaken by on-site readers (assessing participants at their own site) and during central reading sessions by 3 independent, blinded readers.
Time Frame: Unenhanced MRI: Baseline Period (Day -1 to Day 0); mangoral-enhanced MRI: 4 hours after mangoral administration on Day 0; and combined MRI: Baseline Period (Day -1 to Day 0) and 4 hours after mangoral administration on Day 0
Population: FAS: All participants of the Safety Population who received the IMP and for whom the primary efficacy variable was assessable, i.e. all unenhanced / enhanced liver MRI images are assessable.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Mangoral-enhanced MRI: All participants undertook an unenhanced MRI examination of the liver during the Baseline Period (Day -1 to Day 0, i.e., within 24 hours of mangoral administration).
  On the day of MRI (Day 0), all participants received a single oral dose of mangoral (800 mg) after a fast of at least 4 hours and undertook a mangoral-enhanced MRI examination of the liver 4 [±1] hours after mangoral administration.
  Mangoral-enhanced MRI was defined as the reading of the mangoral enhanced MRI only.
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI | Combined MRI
Number analyzed (Participants) | 85 | 85 | 85
lesions
  On-site Readers | 5.7 (9.07) | 6.2 (9.35) | 6.4 (9.57)
  Reader 1: number analyzed (Participants) | 85 | 85 | 84
  Reader 1 | 3.5 (5.18) | 4.3 (5.39) | 4.2 (5.19)
  Reader 2: number analyzed (Participants) | 85 | 85 | 84
  Reader 2 | 3.1 (5.07) | 3.6 (5.34) | 3.2 (4.85)
  Reader 3 | 4.1 (5.58) | 4.5 (5.55) | 4.3 (5.59)

4. Secondary Outcome: Lesion Border Delineation in Mangoral-enhanced MRI Compared to Unenhanced MRI
Description: Visualization of focal liver lesions was measured by variables: 'lesion border delineation' and 'lesion contrast' compared to liver background. Qualitative assessment determined on the 4-point scales for up to 15 lesions per participant. Each lesion was assessed for lesion border delineation from 1 (poor: lesion border is poorly distinct) to 4 (excellent: lesion border is sharply and clearly distinct). Central reading sessions were undertaken by 3 independent, blinded readers.
  The scores were calculated for each participant by summing the individual lesion scores and calculating the mean. The total score could range from 1 to 4 for each participant with higher scores representing a better outcome.
Time Frame: Unenhanced MRI: Baseline Period (Day -1 to Day 0); mangoral-enhanced MRI: 4 hours after mangoral administration on Day 0
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI
Number analyzed (Participants) | 85 | 85
score on a scale
  Reader 1: number analyzed (Participants) | 60 | 60
  Reader 1 | 2.57 (0.783) | 3.34 (0.814)
  Reader 2: number analyzed (Participants) | 52 | 52
  Reader 2 | 2.95 (0.986) | 3.71 (0.647)
  Reader 3: number analyzed (Participants) | 59 | 59
  Reader 3 | 2.27 (0.854) | 2.86 (0.881)
Statistical Analysis 1: Comparison: Unenhanced MRI vs Mangoral-enhanced MRI; Paired difference of mangoral-enhanced MRI versus unenhanced MRI: Reader 1; Test type: Superiority — Reader success was achieved if the reading results demonstrated superiority of mangoral-enhanced MRI versus unenhanced MRI for both lesion border delineation and lesion contrast. The acceptance by two out of three readers was considered to be a successful demonstration of efficacy in the study; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [0.555 to 0.971], Standard Deviation 0.805 — Positive changes in lesion border delineation mean difference (mangoral-enhanced MRI compared to unenhanced MRI) represents a better outcome
Statistical Analysis 2: Comparison: Unenhanced MRI vs Mangoral-enhanced MRI; Paired difference of mangoral-enhanced MRI versus unenhanced MRI: Reader 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [0.464 to 1.054], Standard Deviation 1.059 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Unenhanced MRI vs Mangoral-enhanced MRI; Paired difference of mangoral-enhanced MRI versus unenhanced MRI: Reader 3; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.429 to 0.747], Standard Deviation 0.609 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Lesion Contrast in Mangoral-enhanced MRI Compared to Unenhanced MRI
Description: Visualization of focal liver lesions was measured by variables: 'lesion border delineation' and 'lesion contrast' compared to liver background. Qualitative assessment determined on the 4-point scales for up to 15 lesions per participant. Each lesion was assessed for lesion contrast from 1 (poor: difference in signal intensity between the lesion and the surrounding normal liver tissue is poor) to 4 (excellent: difference in signal intensity between the lesion and the surrounding liver is marked). Central reading sessions were undertaken by 3 independent, blinded readers.
  The scores were calculated for each participant by summing the individual lesion scores and calculating the mean. The total score could range from 1 to 4 for each participant with higher scores representing a better outcome.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI
Number analyzed (Participants) | 85 | 85
score on a scale
  Reader 1: number analyzed (Participants) | 60 | 60
  Reader 1 | 2.57 (0.787) | 3.52 (0.735)
  Reader 2: number analyzed (Participants) | 52 | 52
  Reader 2 | 2.80 (0.940) | 3.53 (0.816)
  Reader 3: number analyzed (Participants) | 59 | 59
  Reader 3 | 2.46 (0.933) | 3.18 (0.882)
Statistical Analysis 1: Comparison: Unenhanced MRI vs Mangoral-enhanced MRI; Paired difference of mangoral-enhanced MRI versus unenhanced MRI: Reader 1; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [0.726 to 1.166], Standard Deviation 0.852 — Positive changes in lesion contrast mean difference (mangoral-enhanced MRI compared to unenhanced MRI) represents a better outcome
Statistical Analysis 2: Comparison: Unenhanced MRI vs Mangoral-enhanced MRI; Paired difference of mangoral-enhanced MRI versus unenhanced MRI: Reader 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [0.380 to 1.082], Standard Deviation 1.261 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Unenhanced MRI vs Mangoral-enhanced MRI; Paired difference of mangoral-enhanced MRI versus unenhanced MRI: Reader 3; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-test, 1 sided; p-values show a one-sided t-test with a significance level of 0.025; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [0.517 to 0.927], Standard Deviation 0.786 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Confidence in Lesion Detection Score
Description: Each lesion was evaluated on a 3-point scale: 1 (lesion is detected with low confidence), 2 (lesion is detected with moderate confidence), 3 (lesion is detected with high confidence). Higher confidence in lesion detection scores represent better outcomes.
  Assessments of unenhanced MRI, mangoral-enhanced MRI, and combined MRI for confidence in lesion detection were undertaken by on-site readers (assessing participants are their own site) and during central reading sessions by 3 independent, blinded readers.
Time Frame: as for outcome 3
Population: FAS: All participants of the Safety Population who received the IMP and for whom the primary efficacy variable was assessable, i.e. all unenhanced / enhanced liver MRI images are assessable. The number of participants analyzed represents the number of participants with analyzed MRI images. Independent readers analyzed a maximum of 15 lesions per participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Lesions
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI | Combined MRI
Number analyzed (Participants) | 85 | 85 | 85
Number analyzed (Lesions) | 387 | 417 | 397
score on a scale
  On-site Readers | 2.5 (0.66) | 2.8 (0.42) | 2.8 (0.47)
  Reader 1: number analyzed (Lesions) | 301 | 362 | 350
  Reader 1 | 2.8 (0.54) | 2.8 (0.53) | 2.8 (0.57)
  Reader 2: number analyzed (Lesions) | 265 | 306 | 265
  Reader 2 | 3.0 (0.26) | 3.0 (0.20) | 2.9 (0.29)
  Reader 3: number analyzed (Lesions) | 347 | 381 | 368
  Reader 3 | 2.8 (0.59) | 2.9 (0.45) | 2.9 (0.38)

7. Secondary Outcome: Confidence in Lesion Localization Score
Description: Each lesion was evaluated on a 3-point scale: 1 (lesion is localized to a liver segment with low confidence), 2 (lesion is localized to a liver segment with moderate confidence), 3 (lesion is localized to a liver segment with high confidence).
  Assessments of unenhanced MRI, mangoral-enhanced MRI, and combined MRI for confidence in lesion localization were undertaken by on-site readers (assessing participants at their own site) and during central reading sessions by 3 independent, blinded readers.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Lesions
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI | Combined MRI
Number analyzed (Participants) | 85 | 85 | 85
Number analyzed (Lesions) | 387 | 417 | 397
score on a scale
  On-site Readers | 2.5 (0.65) | 2.9 (0.42) | 2.8 (0.49)
  Reader 1: number analyzed (Lesions) | 301 | 362 | 350
  Reader 1 | 2.7 (0.57) | 2.8 (0.51) | 2.8 (0.51)
  Reader 2: number analyzed (Lesions) | 265 | 306 | 265
  Reader 2 | 2.9 (0.30) | 3.0 (0.20) | 3.0 (0.19)
  Reader 3: number analyzed (Lesions) | 347 | 381 | 368
  Reader 3 | 2.9 (0.33) | 2.9 (0.26) | 3.0 (0.17)

8. Secondary Outcome: Longest Diameter of Largest and Smallest Lesion
Description: Assessments of unenhanced MRI and mangoral-enhanced MRI for lesion dimensions were undertaken during central reading sessions by 3 independent, blinded readers.
Time Frame: as for outcome 4
Population: FAS: All participants of the Safety Population who received the IMP and for whom the primary efficacy variable was assessable, i.e. all unenhanced / enhanced liver MRI images are assessable. The overall number of participants analyzed includes all participants that contributed data for the outcome measure. The number of participants analyzed per row includes only participants with detected and scored lesions by each reader.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI
Number analyzed (Participants) | 85 | 85
mm
  Smallest Lesion: Reader 1: number analyzed (Participants) | 63 | 69
  Smallest Lesion: Reader 1 | 23.5 (23.75) | 21.4 (24.20)
  Smallest Lesion: Reader 2: number analyzed (Participants) | 57 | 62
  Smallest Lesion: Reader 2 | 27.2 (25.50) | 25.3 (26.46)
  Smallest Lesion: Reader 3: number analyzed (Participants) | 66 | 66
  Smallest Lesion: Reader 3 | 19.8 (23.89) | 17.0 (23.06)
  Largest Lesion: Reader 1: number analyzed (Participants) | 63 | 69
  Largest Lesion: Reader 1 | 42.2 (32.49) | 38.2 (29.53)
  Largest Lesion: Reader 2: number analyzed (Participants) | 57 | 62
  Largest Lesion: Reader 2 | 44.5 (31.49) | 47.9 (36.03)
  Largest Lesion: Reader 3: number analyzed (Participants) | 66 | 66
  Largest Lesion: Reader 3 | 35.5 (31.25) | 35.2 (27.45)

9. Secondary Outcome: Percentage Liver Signal Intensity (SI) Enhancement in Mangoral-enhanced MRI Compared to Unenhanced MRI
Description: Quantitative SI was measured by positioning circular regions of interest in a homogenous area in the liver and the assessed liver lesion on the same image. SI liver was defined as the SI of the liver. Liver SI enhancement (%) = ([SI liver post contrast - SI liver pre contrast] / [SI liver pre contrast]) × 100.
  Assessments of unenhanced MRI and mangoral-enhanced MRI for liver SI were undertaken during central reading sessions by the 3 independent, blinded readers.
Time Frame: as for outcome 4
Population: FAS: All participants of the Safety Population who received the IMP and for whom the primary efficacy variable was assessable, i.e. all unenhanced / enhanced liver MRI images are assessable. As pre-specified in the statistical analysis plan, results are presented for SI enhancement following mangoral-enhanced MRI compared to unenhanced MRI.
Measure: Mean (Standard Deviation); unit: Percentage SI enhancement
Groups:
- Unenhanced MRI and Mangoral-enhanced MRI: All participants undertook an unenhanced MRI examination of the liver during the Baseline Period (Day -1 to Day 0, i.e., within 24 hours of mangoral administration).
  On the day of MRI (Day 0), all participants received a single oral dose of mangoral (800 mg) after a fast of at least 4 hours and undertook a mangoral-enhanced MRI examination of the liver 4 [±1] hours after mangoral administration.
  Mangoral-enhanced MRI was defined as the reading of the mangoral enhanced MRI only.
Arm/Group | Unenhanced MRI and Mangoral-enhanced MRI
Number analyzed (Participants) | 85
Percentage SI enhancement
  Reader 1: number analyzed (Participants) | 73
  Reader 1 | 72.159 (148.2818)
  Reader 2: number analyzed (Participants) | 83
  Reader 2 | 59.633 (113.7548)
  Reader 3 | 61.456 (105.3634)

10. Secondary Outcome: Liver-to-lesion Contrast (LLC) in Mangoral-enhanced MRI Compared to Unenhanced MRI
Description: Quantitative SI was measured by positioning circular regions of interest in a homogenous area in the liver and the assessed liver lesion on the same image. Up to 5 lesions per participant of ≥ 2 cm in diameter were evaluated and these lesions were the same on pre-and post-contrast images. SI lesion was defined as the SI of these lesions. SI liver was defined as the SI of the liver. LLC = (SI liver - SI lesion) / (SI liver + SI lesion). Higher ratio scores represent a better outcome.
  Assessments of unenhanced MRI and mangoral-enhanced MRI for LLC ratio were undertaken during central reading sessions by the 3 independent, blinded readers.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI
Number analyzed (Participants) | 85 | 85
ratio
  Reader 1: number analyzed (Participants) | 70 | 70
  Reader 1 | 0.143 (0.1694) | 0.306 (0.1816)
  Reader 2: number analyzed (Participants) | 57 | 56
  Reader 2 | 0.109 (0.2739) | 0.291 (0.2709)
  Reader 3: number analyzed (Participants) | 47 | 47
  Reader 3 | 0.142 (0.1882) | 0.331 (0.2162)

11. Secondary Outcome: Signal-to-noise Ratio (SNR) in Mangoral-enhanced MRI Compared to Unenhanced MRI
Description: Quantitative SI was measured by positioning circular regions of interest in a homogenous area in the liver and the assessed liver lesion on the same image. SI liver was defined as the SI of the liver. Standard deviation of the background noise was measured using the largest possible rectangular region of interest vertical to the patient's abdomen in the direction of the phase-encoding gradient. SNR = SI liver / standard deviation noise. Higher ratio scores represent a better outcome.
  Assessments of unenhanced MRI and mangoral-enhanced MRI for SNR were undertaken during central reading sessions by the 3 independent, blinded readers.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI
Number analyzed (Participants) | 85 | 85
ratio
  Reader 1: number analyzed (Participants) | 70 | 71
  Reader 1 | 286.428 (581.8717) | 322.951 (365.1663)
  Reader 2: number analyzed (Participants) | 78 | 79
  Reader 2 | 226.367 (362.3748) | 531.223 (1175.7566)
  Reader 3: number analyzed (Participants) | 75 | 79
  Reader 3 | 248.653 (508.6403) | 419.706 (694.8662)

12. Secondary Outcome: Contrast-to-noise Ratio (CNR) in Mangoral-enhanced MRI Compared to Unenhanced MRI
Description: Quantitative SI was measured by positioning circular regions of interest in a homogenous area in the liver and the assessed liver lesion on the same image. Up to 5 lesions per participant of ≥ 2 cm in diameter were evaluated and these lesions were the same on pre-and post-contrast images. SI lesion was defined as the SI of these lesions. SI liver was defined as the SI of the liver. Standard deviation of the background noise was measured using the largest possible rectangular region of interest vertical to the patient's abdomen in the direction of the phase-encoding gradient. CNR = (SI liver - mean of SI lesion) / standard deviation noise. Higher ratio scores represent a better outcome.
  Assessments of unenhanced MRI and mangoral-enhanced MRI for CNR were undertaken during central reading sessions by the 3 independent, blinded readers.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Unenhanced MRI | Mangoral-enhanced MRI
Number analyzed (Participants) | 85 | 85
ratio
  Reader 1: number analyzed (Participants) | 67 | 68
  Reader 1 | 56.564 (197.1474) | 137.281 (161.1640)
  Reader 2: number analyzed (Participants) | 53 | 54
  Reader 2 | 33.506 (214.2616) | 277.270 (650.8484)
  Reader 3: number analyzed (Participants) | 43 | 43
  Reader 3 | 91.019 (306.2666) | 241.093 (510.3520)

13. Secondary Outcome: Number of Participants With Change(s) in Recommended Management Based on Diagnostic Performance of Combined MRI or Mangoral-enhanced MRI Compared to Unenhanced MRI
Description: A participant was considered to have a change in recommended management when compared to unenhanced MRI if recommended management was different following assessment of the combined MRI or mangoral-enhanced MRI, including next steps in management (i.e. chemotherapy, surgery, local ablation procedure, combination therapy, or other [specify]). Recommended patient management from "other" in unenhanced MRI to "other" in combined MRI or mangoral-enhanced MRI was considered not a change regardless of the free text.
  Assessments of unenhanced MRI, mangoral-enhanced MRI, and combined MRI for confidence in lesion detection were undertaken by on-site readers (assessing participants at their own site with access to patient records) and during central reading sessions by 3 independent, blinded readers (without access to patient records).
Time Frame: as for outcome 3
Population: FAS: All participants of the Safety Population who received the IMP and for whom the primary efficacy variable was assessable, i.e. all unenhanced / enhanced liver MRI images are assessable. As pre-specified in the statistical analysis plan, results are presented for change in recommended management following combined MRI and mangoral-enhanced MRI only.
Measure: Count of Participants; unit: Participants
Arm/Group | Mangoral-enhanced MRI | Combined MRI
Number analyzed (Participants) | 85 | 85
Participants
  On-site Readers: number analyzed (Participants) | 83 | 83
  On-site Readers | 4 | 4
  Reader 1: number analyzed (Participants) | 85 | 84
  Reader 1 | 19 | 21
  Reader 2: number analyzed (Participants) | 85 | 84
  Reader 2 | 27 | 29
  Reader 3 | 19 | 19

ADVERSE EVENTS:
Time Frame: Up to Day 7
Description: Safety Population: All participants enrolled in the study (fulfil all inclusion criteria, but none of the exclusion criteria and have been included in the clinical study at Visit 2).
Arm/Group | Mangoral
All-Cause Mortality (participants affected / at risk) | 1/87
Serious Adverse Events (participants affected / at risk) | 2/87
Other Adverse Events (participants affected / at risk) | 41/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mangoral (N=87)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mangoral (N=87)
Nausea (Gastrointestinal disorders) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 12 (13)
Vomiting (Gastrointestinal disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Retching (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Blood urea increased (Investigations) | 3 (7)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
Neutrophil count increased (Investigations) | 1 (1)
White blood cells urine positive (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatine increased (Investigations) | 1 (5)
Blood creatinine increased (Investigations) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood pressure systolic increased (Investigations) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT04119843/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT04119843/SAP_001.pdf